CLINICAL TRIAL: NCT04351711
Title: Immunological Profiling of Patients With COVID-19 in Respiratory Distress
Acronym: ACTICOV-2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Institute of Human Genetics, Montpellier (Unknown)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2020-01/PC-01; 2020-A00875-34 (Other: ANSM)
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: SARS-CoV-2; Covid-19
Keywords: respiratory failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and peripheral blood mononuclear cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Patients SARS-CoV-2 with respiratory failure: Patients in intensive care
  Interventions: Other: Immunological profiling
- Patients SARS-CoV-2 without respiratory failure: Patients hospitalized in normal hospital wards
  Interventions: Other: Immunological profiling
- HEALTHY VOLUNTEERS: HEALTHY VOLUNTEERS
  Interventions: Other: Immunological profiling
- NON-COVID-19 PATIENTS: Patient hospitalized at the CHU of Nîmes for an infection by a virus other than SARS-CoV-2
  Interventions: Other: Immunological profiling
- PAUCISYMPTOMATIC SARS-COV-2+ PATIENTS: Patient positive for SARS-CoV-2 by RT-PCR at the CHU of Nîmes and presenting at most moderate clinical signs without respiratory insufficiency (O2 saturation greater than or equal to 96%) during the confinement period
  Interventions: Other: Immunological profiling
- convalescent patients: Additional 1-year follow-up visit
  Interventions: Other: Immunological profiling

INTERVENTIONS:
Other: Immunological profiling — The immune activation phenotype will be assessed using a standardized panel of soluble and membrane immune activation markers
Other: Immunological profiling — The immune activation phenotype will be assessed using a standardized panel of soluble and membrane immune activation markers
  Other Names: Additional 1-year follow-up visit for 30 convalescent patients
  Groups: convalescent patients

SUMMARY:
The study investigators hypothesize that the pneumonia arising in patients with COVID-19 is largely of immunopathological origin. The investigators will therefore seek to define the immune activation phenotype of patients in respiratory distress and to see if this immune signature is predictive of mortality. Finally, the investigators will look for overproduced inflammatory mediators to identify potential therapeutic targets.

DETAILED DESCRIPTION:
SARS-CoV inhibits the viral detection systems and the signaling pathways of type I interferons (IFN-I). The weakness of the initial interferon response is predictive of the severity of future lung disease. The effectiveness of this escape strategy seems to allow these coronaviruses to replicate in the human body without triggering an effective innate immune response. This could explain the contagiousness of asymptomatic infected people.

However, this initial replication causes a cytokine storm involving inflammatory cytokines. The intensity of this cytokine storm is correlated with the severity of COVID-19 cases.

Pulmonary involvement, which is the main cause of death in SARS-CoV infections, has been attributed to local inflammation, with infiltration of CD8 + T cells, polymorphonuclear cells, monocytes and macrophages, infiltration proportional to the severity of respiratory failure as well as increased vascular permeability.

SARS-CoV also induces T cell apoptosis. This pro-apoptotic effect could contribute to the lymphopenia observed in 37 to 63% of COVID-19 cases, which is predictive of severe forms.

Thus the pulmonary involvement could be partly caused by immunopathological mechanisms.

Immunological disturbances associated with respiratory failure need to be better defined. Recently, we measured a panel of soluble and membrane markers allowing to characterize T CD4 +, T CD8 +, B, monocytic, NK, endothelial activation as well as inflammation in a sample made up of 150 volunteers from a general population providing a control population.

The study investigators aim to use this panel to define the immune activation state of patients infected with SARS-CoV-2 hospitalized for respiratory distress. In addition, the investigators will identify the soluble factors linked to the immune activation overproduced by the peripheral blood mononuclear cells (PBMC) of these patients. Finally, the investigators want to characterize the transcriptome of the main circulating immune sub-populations. These parameters will be compared with those of patients infected with SARS-CoV-2 hospitalized before experiencing respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be a member or beneficiary of a health insurance plan
* Patient hospitalized in respiratory resuscitation or in the service of Infectious and Tropical Diseases of the CHU de Nîmes with infection by SARS-CoV-2, confirmed by RT-PCR or by an antigen test.

Exclusion Criteria:

* The subject is in a period of exclusion determined by a previous study
* The patient is under safeguard of justice
* Patient already under ventilation transferred from another center

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in intensive care or normal hospitalization at the CHU de Nîmes for SARS-CoV-2 infection, confirmed by PT-PCR or by an antigen test
  Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Membrane expression of Human Leukocyte Antigen -DR isotype compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Membrane expression of cluster of differentiation 38 compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Membrane expression of Programmed cell death 1 protein compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Membrane expression of cluster of differentiation 45RA compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry
Membrane expression of cluster of differentiation 27 (naïve/central memory/effector memory) compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Membrane expression of CD57 on T CD4+ and T CD8+ cells compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Membrane expression of cluster of differentiation 27 on T CD4+ and T CD8+ cells compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Membrane expression of cluster of differentiation 28 on T CD4+ and T CD8+ cells compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Membrane expression of Human Leukocyte Antigen -DR isotype on Naturel Killer cells compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Membrane expression of cluster of differentiation 69 on Naturel Killer cells compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Membrane expression of cluster of differentiation 56 on Naturel Killer cells compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Membrane expression of cluster of differentiation 57 on Naturel Killer cells compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Membrane expression of cluster of differentiation 14 on Naturel Killer cells compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Membrane expression of cluster of differentiation 16 on Naturel Killer cells compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Number of regulatory T cells (CD4+CD25hiCD127loFoxP3+). | Day 0
  Quantified by flow cytometry; % variation / normal values
Percentage of regulatory T cells (CD4+CD25hiCD127loFoxP3+). | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Immunoglobulin A compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Immunoglobulin G compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Immunoglobulin M compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Soluble cluster of differentiation 14 compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Soluble cluster of differentiation 163 compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Ultrasensitive C-Reactive Protein compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Soluble tumor necrosis factor alpha receptor type I compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating E-selectin (cluster of differentiation 62E) compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Granulocyte Macrophage Colony-Stimulating Factor compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry
Rate of circulating InterCellular Adhesion Molecule-1 compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Interferon alpha compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Interferon beta compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Interferon gamma compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Interleukin-1 alpha compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Interleukin-1 beta compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Interleukin-4 compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Interleukin-6 compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Interleukin-8 compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Interleukin-10 compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Interleukin-12p70 compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry
Rate of circulating Interleukin-13 compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Interleukin-17A compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Induced Protein 10 (C-X-C motif chemokine 10) compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Monocyte Chemoattractant Protein-1 (C-C Motif Chemokine Ligand 2) compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Macrophage inflammatory protein-1 alpha (C-C Motif Chemokine Ligand 3) compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating Macrophage inflammatory protein-1 beta (C-C Motif Chemokine Ligand 4) compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of circulating P-selectin compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of tumor necrosis factor alpha compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of tissue plasminogen activator compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of soluble form of endothelial protein C receptor compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values
Rate of D-Dimers compared to normal values (based on 150 healthy volunteers previously sampled) | Day 0
  Quantified by flow cytometry; % variation / normal values

SECONDARY OUTCOMES:
Compare the immune activation phenotype (defined in primary outcome) of patients affected by COVID-19 before any respiratory distress against that of 150 volunteers from the general population (data already existing). | Day 0
  Difference in expression of the biomarkers assayed for primary outcome
Compare the immune activation phenotype (defined in primary outcome) of patients affected by COVID-19 with respiratory failure against versus those without respiratory failure | Day 0
  Difference in expression of the biomarkers assayed for primary outcome
Mortality rate | End of study (2021)
  Mortality
Comparison of E-selectin levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Granulocyte Macrophage Colony-Stimulating Factor levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of InterCellular Adhesion Molecule levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Interferon alpha levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Interferon gamma levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Interleukin-1alpha levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Interleukin-1beta levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Interleukin-4 levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Interleukin-6 levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Interleukin-8 (C-X-C motif ligand 8) levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Interleukin-10 levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Interleukin-12p70 levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Interleukin-13 levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Interleukin-17A levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Induced Protein -10 (C-X-C motif chemokine 10) levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Monocyte Chemoattractant Protein-1 levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Macrophage Inflammatory Protein-1alpha levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Macrophage Inflammatory Protein -1beta levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of P-Selectin levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Comparison of Tumor necrosis factor alpha levels from plasma and the supernatant of PBMC activated or not by lipopolysaccharide and Staphylococcal enterotoxin B against norms previously established from 16 healthy subjects | Day 0
  quantified by Luminex (TruCulture tube system (Myriad RBM))
Identify inflammatory mediators over-produced by the PBMC of patients with COVID-19 before respiratory distress | Day 0
  Difference in expression of the 20 inflammatory markers described in outcomes 51-70
Compare the inflammatory mediators over-produced by the peripheral blood mononuclear cells of patients with COVID-19 with versus without respiratory failure | Day 0
  Difference in expression of the 20 inflammatory markers described in outcomes 51-70
Comparison of transcriptome from peripheral blood mononuclear cells from 12 patients with respiratory failure (from intensive care ward) and 10 without (normal hospitalization) | Day 0
  Performed at the Institut de Génétique Humaine (Montpellier)
To evaluate whether lymphocyte apoptosis measured in the acute phase is predictive of residual specific Ac levels and B and T immune memory one year later. | 1 year
  Lymphocyte caspase activity
o evaluate whether lymphocyte apoptosis measured in the acute phase is predictive of residual specific Ac levels and B and T immune memory one year later. | 1 year
  circulating FasL level
o evaluate whether lymphocyte apoptosis measured in the acute phase is predictive of residual specific Ac levels and B and T immune memory one year later. | 1 year
  expression of phosphatidylserine on the surface of lymphocytes in the acute phase
o evaluate whether lymphocyte apoptosis measured in the acute phase is predictive of residual specific Ac levels and B and T immune memory one year later. | 1 year
  levels of Ac
o evaluate whether lymphocyte apoptosis measured in the acute phase is predictive of residual specific Ac levels and B and T immune memory one year later. | 1 year
  plasmablasts and specific T cells

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Corbeau, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France

REFERENCES:
- [Result] Andre S, Picard M, Cezar R, Roux-Dalvai F, Alleaume-Butaux A, Soundaramourty C, Cruz AS, Mendes-Frias A, Gotti C, Leclercq M, Nicolas A, Tauzin A, Carvalho A, Capela C, Pedrosa J, Castro AG, Kundura L, Loubet P, Sotto A, Muller L, Lefrant JY, Roger C, Claret PG, Duvnjak S, Tran TA, Racine G, Zghidi-Abouzid O, Nioche P, Silvestre R, Droit A, Mammano F, Corbeau P, Estaquier J. T cell apoptosis characterizes severe Covid-19 disease. Cell Death Differ. 2022 Aug;29(8):1486-1499. doi: 10.1038/s41418-022-00936-x. Epub 2022 Jan 22. PMID 35066575